CLINICAL TRIAL: NCT02802124
Title: Phase I Trial Evaluating Carbon Ion Radiotherapy for the Treatment of Chinese Hepatocellular Carcinoma
Brief Title: Carbon Ion Radiotherapy for the Treatment of Chinese Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For tumor locates away from GI the planned enrolled patient had been completed, but for tumor locates closely to GI only 6 patients had been enrolled because not many eligible patients were available.
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Guoliang Jiang, Director the committee of clinical technique, Shanghai Proton and Heavy Ion Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HCC2016-01
Record Dates: First submitted 2016-06-12; First posted 2016-06-16 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; carbon-ion radiotherapy; toxicity; efficacy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carbon-ion radiotherapy for tumor away from GI (Experimental): For tumor location which is away from gastrointestine (the distance is more than 1 cm). We use carbon-ion radiotherapy for the treatment of hepatocellular carcinoma. Four dose levels [55 Gray equivalent (GyE)/10 fractions (Fx), 60GyE/10Fx, 65GyE/10Fx, 70GyE/10Fx] are planned within the Phase I part.
  Interventions: Radiation: carbon-ion radiotherapy for tumor away from GI
- carbon-ion radiotherapy for tumor adjacent to GI (Experimental): For tumor location which is adjacent to gastrointestine (less than 1 cm).We use carbon-ion radiotherapy for the treatment of hepatocellular carcinoma.
  Three dose levels (carbon 60GyE/15Fx, carbon 67.5GyE/15Fx, carbon 75GyE/15Fx) are planned within the Phase I part.
  Interventions: Radiation: carbon-ion radiotherapy for tumor adjacent to GI

INTERVENTIONS:
Radiation: carbon-ion radiotherapy for tumor away from GI
  Arms: carbon-ion radiotherapy for tumor away from GI
Radiation: carbon-ion radiotherapy for tumor adjacent to GI
  Arms: carbon-ion radiotherapy for tumor adjacent to GI

SUMMARY:
The aim of this research project is to assess the feasibility and safety of carbon-ion radiotherapy for the treatment of localized Chinese hepatocellular carcinoma

DETAILED DESCRIPTION:
The purpose of this study is to determine the maximal tolerated dose (MTD) of carbon ion radiotherapy (CIRT) in the treatment of localized Chinese hepatocellular carcinoma with respective to toxicity and tumor control. Participants will be treated with CIRT with escalating dose regimens based on the tumor location to evaluate the maximal tolerated dose (MTD) in terms of acute and subacute toxicity observed during and within 3 months after the completion of CIRT. Primary endpoint is toxicity, second endpoint is progression-free survival, overall survival and tumor response.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed hepatocellular carcinoma (HCC) or clinical diagnosis of HCC according to American association for the study of liver diseases （AASLD）-guidelines or clinical diagnosis criteria based on Alpha Fetoprotein （AFP), and radiological images proposed by Liver Cancer Society, Chinese Anti-Cancer Association;
2. no clinically distant metastasis;
3. Child Push score A,technically unresectable, or medically inoperable; maximal tumor size is less than 12 cm;
4. age ≥ 18 and <80 years of age;
5. Karnofsky Performance Score ≥ 70;
6. No previous invasive cancer (within 5 years before the HCC diagnosis)except for skin non-melanoma cancer or non muscle invasive bladder cancer; Ability to understand character and individual consequences of the clinical trial;
7. Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial;

Exclusion Criteria:

1. Distant metastasis (M1);
2. maximal tumor size is more than 12 cm;
3. tumor invading adjacent gastrointestine (T4);
4. Child push score B or C;
5. Previous hepatic radiotherapy;
6. Severe systemic disorders;
7. Previous malignancy (within 5 years) except for skin non-melanoma cancer or 3-year disease free interval from previous malignancy like in situ cervix cancer or non muscle invasive bladder cancer;
8. Non conformity of the radiotherapy dose distribution when compared to the dose constraints;
9. Psychiatric disorders or any other condition that can make unreliable the informed consent;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2023-10 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Time interval from the start of CIRT to 3 months after the completion of CIRT
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Overall survival of all patients | From the diagnosis of localized hepatocellular carcinoma, a median of 2 years
  Overall survival of all patients
Progression-free survival of all patients | From the diagnosis of localized hepatocellular carcinoma, a median of 2 years
  Progression-free survival of all patients
Number of participants with tumor response as assessed by RECIST 1.1 | Time interval from the start of CIRT to 3 months after the completion of CIRT
  Number of participants with tumor response as assessed by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: guoliang Jiang, Prof., Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No